CLINICAL TRIAL: NCT03630679
Title: A Pilot Study Evaluating Sleep, Stress, and Infant Nutrition Using a Chatbot With Parents of Preterm and Full-term Infants
Brief Title: A Study Evaluating Sleep, Stress and Infant Nutrition Using a Chatbot
Status: Completed | Type: Observational
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Collaborators: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: OBVIO-DAN-003
Record Dates: First submitted 2018-07-17; First posted 2018-08-15 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Preterm Birth; Healthy
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm: born at <37 weeks of gestation
- Full term Term: born at >/= 37 weeks of gestation

SUMMARY:
20 parents with healthy preterm infants (born at <37 weeks of gestation), age 0-6 months and discharged from the hospital at time of enrollment and 20 parents with healthy full-term infants (born at ≥37 weeks of gestation), age 0-6 months and discharged from the hospital at time of enrollment will be enrolled to obtain records of sleep, stress, and infant nutrition from parents of infants (preterm and full-term) through interaction with the study chatbot.

DETAILED DESCRIPTION:
20 parents with healthy preterm infants (born at <37 weeks of gestation), age 0-6 months and discharged from the hospital at time of enrollment and 20 parents with healthy full-term infants (born at ≥37 weeks of gestation), age 0-6 months and discharged from the hospital at time of enrollment will be enrolled to obtain records of sleep, stress, and infant nutrition from parents of infants (preterm and full-term) through interaction with the study chatbot.

Data obtained from parents of preterm infants and parents of full-term infants on sleep, stress, and infant nutrition will be compared.

An evaluation of the usability of the mobile app hosting the chatbot, the study chatbot and its functionality in general among this population will also be conducted

ELIGIBILITY:
Inclusion Criteria:

Subjects (parent and infant) must meet the following criteria:

* Healthy infants (preterm and full-term) must be 0-6 months of age at time of enrollment
* Infants must be at home (discharged from the hospital) at time of enrollment
* Informed consent from parent whose age is ≥21 years
* Parent must be proficient in the English language
* Parent must be able to comply with the required study tasks, as per PI's judgment
* In-home access to reliable internet connections; a mobile device suitable for electronic communication

Exclusion Criteria:

Infant must not meet any of the following criteria:

* Known to have current or previous illnesses/conditions which could interfere with the study outcome (per PI's clinical judgment)
* Must not be currently participating in any other clinical study

Parent must not meet any of the following criteria:

* Must not be known to have a significant medical condition that might interfere with the study (per PI's clinical judgment) that meets one of the following criteria:
* Presence of current mental illness or history of mental illness
* Any acute or chronic illness that makes the parent unsuitable for the study based on the PI's judgment
* Must not be a single parent
* Inability of the parent to comply with the study protocol or PI's uncertainty about the willingness or ability of the parent to comply with the protocol requirements

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * 20 parents with healthy preterm infants (born at <37 weeks of gestation), age 0-6 months and discharged from the hospital at time of enrollment
  * 20 parents with healthy full-term infants (born at ≥37 weeks of gestation), age 0-6 months and discharged from the hospital at time of enrollment
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mei Chien Chua, MBBS, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong J, Foussat AC, Ting S, Acerbi E, van Elburg RM, Mei Chien C. A Chatbot to Engage Parents of Preterm and Term Infants on Parental Stress, Parental Sleep, and Infant Feeding: Usability and Feasibility Study. JMIR Pediatr Parent. 2021 Oct 26;4(4):e30169. doi: 10.2196/30169. PMID 34544679

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Preterm | Full Term Term
Started | 20 | 25
Completed | 13 | 13
Not Completed | 7 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preterm | Full Term Term | Total
Number analyzed (Participants) | 20 | 25 | 45
Age, Customized [Count of Participants; unit: Participants]
  Parent's age: 21-25 years old | 2 | 1 | 3
  Parent's age: 26-30 years old | 3 | 10 | 13
  Parent's age: 31-35 years old | 10 | 8 | 18
  Parent's age: 36-40 years old | 4 | 6 | 10
  Parent's age: 41-45 years old | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 10 | 12 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Singapore | 20 | 25 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Chats on Sleep, Stress and Infant Nutrition
Description: Obtaining number of chats for sleep, stress, and infant nutrition from parents of infants (preterm and full-term) through interaction with the study chatbot
Time Frame: 8 weeks
Measure: Number; unit: Chats
Arm/Group | Preterm | Full Term Term
Number analyzed (Participants) | 20 | 25
Chats | 131 | 125

2. Secondary Outcome: Ratings by Parents of Quality of Their Sleep
Description: Comparison on ratings for quality of their (parent) sleep from parents of preterm infants and parents of full-term infants
Time Frame: 8 weeks
Population: Per Protocol
Measure: Number; unit: chat responses
Arm/Group | Preterm | Full Term Term
Number analyzed (Participants) | 13 | 13
chat responses
  1 (Very Good) | 20 | 13
  2 (Good) | 42 | 48
  3 (Bad) | 55 | 38
  4 (Very Bad) | 5 | 7

3. Secondary Outcome: Particular Reasons for Stress Caused by the Baby
Description: Comparison of particular reasons for stress caused by the baby from parents of preterm infants and parents of full-term infants
Time Frame: 8 weeks
Population: Per Protocol
Measure: Number; unit: chat responses
Arm/Group | Preterm | Full Term Term
Number analyzed (Participants) | 13 | 13
chat responses
  My baby is crying a lot | 0 | 3
  My baby is sick | 4 | 0
  My baby's feeding habits | 3 | 3
  My baby's growth | 1 | 1
  My baby's sleeping patterns | 0 | 1
  Other | 9 | 0

4. Secondary Outcome: Number of Chats on Feedings Among Parents Who Give Their Infants Formula
Description: Comparison of number of chats on the feeding from parents of preterm infants and parents of full-term infants who give their infants formula
Time Frame: 8 weeks
Population: Per Protocol
Measure: Number; unit: chat responses
Arm/Group | Preterm | Full Term Term
Number analyzed (Participants) | 13 | 13
chat responses
  0 to 3 | 19 | 13
  4 to 7 | 30 | 19
  8 to 11 | 22 | 13
  12 and above | 1 | 1

5. Other Pre Specified Outcome: Satisfaction Scale Scores for Chatbot and ClaimIt
Description: Satisfaction scale scores for Chatbot and ClaimIt based on a scale score of 1 (very dissatisfied) to 5 (very satisfied) on the Usability of Chatbot and ClaimIt eQuestionnaire
Time Frame: 8 weeks
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Preterm | Full Term Term
Number analyzed (Participants) | 13 | 13
score on a scale
  Chatbot Satisfaction | 3.62 (0.96) | 4.0 (0.82)
  ClaimIt Satisfaction | 3.69 (0.85) | 3.92 (0.76)

ADVERSE EVENTS:
Time Frame: duration of the study - 4 months
Arm/Group | Preterm | Full Term Term
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/25
Other Adverse Events (participants affected / at risk) | 0/20 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/79/NCT03630679/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT03630679/SAP_001.pdf